CLINICAL TRIAL: NCT00680537
Title: Physical Therapy Program for Prevention of Shoulder Pain After Device Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UTSW IRB # 082006-080
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Shoulder Pain
Keywords: physical therapy program
MeSH Terms: conditions — Shoulder Pain | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Control group
- 2 (Experimental): Exercise group
  Interventions: Procedure: Exercises

INTERVENTIONS:
Procedure: Exercises — Completion of a series of shoulder exercises for 6 weeks post device implant
  Arms: 2

SUMMARY:
This is a clinical research study to determine if a prescribed physical therapy intervention after subcutaneous implantation of an implanted cardioverter-defibrillator (ICD) or pacemaker reduces the incidence of rotator cuff tendonitis when compared to usual post procedural care.

DETAILED DESCRIPTION:
One hundred patients who undergo subcutaneous ICD or pacemaker implant and consent to inclusion in the trial will be randomized to one of two groups. One group will receive standard of care instructions after implant. These standard instructions include: no pushing or pulling movements with arm on side of implant, no lifting over 5 lbs., and no movements above the level of the shoulder for six weeks post implant. This will be the control group. The second group, the exercise group, will be instructed verbally on a series of specific exercises (appendix A) to be completed at least three days per week for 6 weeks.

After the patient signs informed consent, a demographic form will be completed. At this enrollment visit, both groups will be asked to use a visual analog scale to report level of shoulder and/or extremity discomfort. Physical exam will include the impingement test, assessment of shoulder elevation, and measurement of the angle of abduction at which discomfort occurs. Subjects will be given the QuickDASH questionnaire (Appendix B) to complete. This questionnaire is an 11 item self-report questionnaire designed to assess the physical function and symptoms during certain activities.

At the 1 week follow-up visit, the patient will be informed of their randomization group. The patients in the control group will receive standard of care instructions. The patients in the exercise group will have specific exercises demonstrated to them and written instructions with pictures will be provided for home reference. Follow-up for both groups will occur at 1, 3 and 6 months post implant and it will include a physical exam, the QuickDASH questionnaire, and the visual analog scale. Patients in the exercise group will be asked to complete an exercise log and return it to the study staff after the 6 week of exercise is complete. In addition, telephone follow-ups will be completed for the exercise group at 2, 3, 5, and 6 weeks post implant. Patients will be asked how often they complete the exercises.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing ICD or pacemaker device implant

Exclusion Criteria:

* Prior shoulder injury or surgery
* Mastectomy on affected side
* CVA with ipsilateral arm involvement
* Inability or refusal to perform exercises as prescribed.
* Subjects who would not be able to come in for follow-up visits at one, three, and six-month intervals will also be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
to determine if a prescribed physical therapy intervention after subcutaneous implantation of an implanted cardioverter-defibrillator (ICD) or pacemaker reduces the incidence of rotator cuff tendonitis when compared to usual post procedural care. | 6 mo

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Joglar, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States